CLINICAL TRIAL: NCT04021576
Title: Fitness- and Health-related Effects of a Sports Injury Prevention Program in Competitive Alpine Skiers
Acronym: ISPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Joerg Spoerri, Principal Investigator, Balgrist University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ISPA
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Athletics

STUDY DESIGN:
Intervention Model Description: Intervention with historical control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): preventative training program
  Interventions: Other: preventative training program
- control (No Intervention): no such training

INTERVENTIONS:
Other: preventative training program — complementary training of leg-, hip- and core-strength/stability
  Arms: intervention

SUMMARY:
Overall Goal: Elaboration of an evidence-based, national prevention strategy to protect the health of competitive alpine skiers, with a particular focus on youth athletes.

Background: Competitive alpine skiing has a relatively high injury risk. 60% of all athletes suffer from a severe knee injury in the early stages of their career, and 20% struggle with recurrent overuse problems of the knee and lower back.

Research Aims: (1) to investigate the effects of a 12-month sports injury prevention program on training attitudes, eccentric hamstring strength, leg axis-/hip-/core-stability and general fitness in competitive alpine skiers; (2) to assess the effectiveness the aforementioned prevention program to lower the occurring health problems in competitive alpine skiers; (3) to identify different pain conditions (knee, back, no pain) based on data measured with smartphones; and (4) to investigate the agreement of self-reported questionnaire data with measured smartphone data and pain as an affecting factor.

Methods: 12-month intervention a sports injury prevention program, a prospective health- and training/activity-monitoring, as well as assessments of eccentric hamstring strength, leg axis/hip/core stability and general fitness at baseline and follow-up.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. to investigate the effects of a sports injury prevention program on train-ing attitudes, eccentric hamstring strength, leg axis-/hip-/core-stability and general fitness in competitive alpine skiers;
2. to assess the effectiveness the prevention program to lower the occur-ring health problems (i.e. traumatic injuries, overuse injuries and illnesses) in competitive alpine skiers.

   The secondary objectives of this study are:
3. to investigate the agreement between self-reported questionnaire data with unobtrusively measured smartphone data (i.e. sensor-based activity data) to monitor the prevention program;
4. to identify athletes at risk for developing pain and injury based on digitally acquired data (questionnaires and activity sensor data).

The primary study outcomes are the changes in training attitudes, maximal eccentric hamstring strength, leg axis-/hip-/core-stability, general fitness-related factors and the occurring health problems in competitive youth alpine skiers over a 12-month intervention period. These outcomes are assessed by established methods of strength testing, neuromuscular screening, and load- and health-monitoring.

The secondary outcome is a smartphone enabled training and injury prevention program for skiing athletes.

Study design: Medical Training Therapy (MTT) Intervention with historical control Group

Methods and procedures:

Fitness- and health-related factors are assessed before and after a 12-month observational period and before and after a 12-month preventative training intervention period.

Maximal eccentric hamstring strength is tested by using the NordBord (Inc. VALD Performance, AU).

Leg axis-/hip-/core-stability related measures are assessed by biomechani-cal measurement technologies, such as Vicon Vero (Inc. Vicon Motion Sys-tems Ltd, UK), mobile 2D force plates (MLD, Inc. SP Sportdiagnosegeräte GmbH, AT), mobile 3D force plates (Inc. Kistler Group, SUI) and surface electromyography (EMG) (aktos, Inc. Myon AG, SUI).

General fitness-related factors are quantified by the Swiss-Ski Power Test (incl. the tasks "swiss cross", "push up", "5-jump", "standing long jump", "twist test", "obstacle course", "high box jump" and "12' run").

The athletes' training loads/activities are monitored using custom question-naires and measurements obtained through a smartphone (i.e. activity sen-sors).

The athletes' health is monitored by the OSTRC questionnaire. The athletes' biological age/maturity offset is estimated according to the non-invasive, anthropometric-based method of Mirwald et al.

Intervention: The intervention (i.e. the preventative training program) includes a specific, complementary training of leg-, hip- and core-strength/stability and will be conducted over an intervention period of 12 months. The control interven-tion, compromises no such training program.

ELIGIBILITY:
Inclusion Criteria:

* competitive athletes that are part of a Swiss-Ski development program
* Written informed consent by the participant (or parents)

Exclusion Criteria:

* No written informed consent

Ages: 13 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 12 months maximal eccentric hamstring strength | assessed before and after a 12-month preventative training intervention
  tested by using the NordBord
Change from baseline to 12 months axis-stability | assessed before and after a 12-month preventative training intervention
  assessed by biomechanical measurement technology
Change from baseline to 12 months hip-stability | assessed before and after a 12-month preventative training intervention
  assessed by biomechanical measurement technology
Change from baseline to 12 months core-stability | assessed before and after a 12-month preventative training intervention
  assessed by biomechanical measurement technology
Change from baseline to 12 months general fitness-related factors | assessed before and after a 12-month preventative training intervention
  quantified by the Swiss-Ski Power Test (incl. the tasks "swiss cross", "push up", "5-jump", "standing long jump", "twist test", "obstacle course", "high box jump" and "12' run")
occurring health problems | 2-weekly
  Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire

SECONDARY OUTCOMES:
smartphone enabled training and injury prevention program | during 12-month preventative training intervention
  senor-based activity measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Spörri, PD Dr., Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital Balgrist Move>Med, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No